CLINICAL TRIAL: NCT06661915
Title: A Randomized Phase 2 Trial of ASTX727 +/- Iadademstat in Accelerated/Blast-Phase Philadelphia Chromosome-Negative Myeloproliferative Neoplasms (MPNs)
Brief Title: A Randomized Study of ASTX727 With or Without Iadademstat in Advanced Myeloproliferative Neoplasms (MPNs)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-08860; NCI-2024-08860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10675 (Other: City of Hope Comprehensive Cancer Center LAO); 10675 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Accelerated Phase Myeloproliferative Neoplasm; Blast Phase Myeloproliferative Neoplasm; Essential Thrombocythemia; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm, Not Otherwise Specified; Polycythemia Vera; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Thrombocythemia, Essential; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis | interventions — Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; iadademstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ASTX727) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo buccal swab sample collection at baseline and blood sample collection and bone marrow aspiration and biopsy throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine
- Arm II (ASTX727, iadademstat) (Experimental): Patients receive ASTX727 PO QD on days 1-5 and iadademstat PO QD on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo buccal swab sample collection at baseline and blood sample collection and bone marrow aspiration and biopsy throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Iadademstat

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo buccal swab and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Iadademstat — Given PO
  Other Names: ORY 1001; ORY-1001; RG 6016; RG6016; RO 7051790; RO7051790; trans-N1-((1R,2S)-2-Phenylcyclopropyl)-1,4-cyclohexanediamine
  Arms: Arm II (ASTX727, iadademstat)

SUMMARY:
This phase II trial compares the effect of ASTX727 in combination with iadademstat to ASTX727 alone in treating patients with accelerated or blast phase Philadelphia chromosome negative myeloproliferative neoplasms (MPNs). ASTX727 is a combination of two drugs, cedazuridine and decitabine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Iadademstat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving ASTX727 in combination with iadademstat may be more effective than ASTX727 alone in treating patients with accelerated or blast phase Philadelphia chromosome negative MPNs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the acute leukemia response-complete (ALR-C) rate of iadademstat + ASTX727 (35 mg decitabine + 100 mg cedazuridine) and ASTX727 (35 mg decitabine + 100 mg cedazuridine) monotherapy within 4 cycles of therapy in patients with accelerated/blast-phase myeloproliferative neoplasms (MPN-AP/BP) previously untreated with deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi).

SECONDARY OBJECTIVE:

I. To compare event-free survival (EFS), overall survival (OS), and percentage of patients going onto allogeneic hematopoietic stem cell transplant (allo-HCT) of iadademstat + ASTX727 (35 mg decitabine + 100 mg cedazuridine) and ASTX727 (35 mg decitabine + 100 mg cedazuridine) monotherapy in patients with MPN-AP/BP previously untreated with DNMTi.

EXPLORATORY OBJECTIVES:

I. To compare iadademstat target engagement between patients treated with iadademstat + ASTX727 (35 mg decitabine + 100 mg cedazuridine) and ASTX727 (35 mg decitabine + 100 mg cedazuridine) monotherapy by evaluating transcriptional changes in proliferative pathways implicated in MPN-AP/BP development and/or progression.

II. To elucidate the common molecular pathways of resistance/progression in patients with MPN-AP/BP receiving DNMTi-based therapy.

III. To measure response using the European LeukemiaNet 2022 Acute Myeloid Leukemia (AML) criteria (Döhner et al., 2022) and compare with the 2012 MPN-BP criteria that is being utilized for primary objective assessment.

OUTLINE: This is a dose escalation study of ASTX727 and iadademstat followed by a randomized study. Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ASTX727 orally (PO) once daily (QD) on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo buccal swab sample collection at baseline and blood sample collection and bone marrow aspiration and biopsy throughout the study.

ARM II: Patients receive ASTX727 PO QD on days 1-5 and iadademstat PO QD on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo buccal swab sample collection at baseline and blood sample collection and bone marrow aspiration and biopsy throughout the study.

After completion of study treatment, patients who stop the study for reasons other than disease progression are followed up every 3 months. Patients who stop the study due to disease progression, are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have morphologically confirmed diagnosis of Philadelphia-chromosome negative MPN in accelerated-phase (10-19% myeloid blasts) or blast-phase (≥ 20% myeloid blasts) arising from polycythemia vera, essential thrombocythemia, primary myelofibrosis, secondary myelofibrosis, or MPN not otherwise specified, as per the World Health Organization (WHO) 2016 classification OR myelodysplastic syndrome (MDS)/MPN overlap syndromes (e.g., chronic myelomonocytic leukemia [CMML]) with ≥ 10% blasts
* Patients must not have received prior DNMTi. Previous use of janus kinase (JAK) inhibition, hydroxyurea, and interferon is allowed. There is no required washout period
* Age ≥ 18 years

  * Because no dosing or adverse event data are currently available on the use of ASTX727 (35 mg decitabine + 100 mg cedazuridine) in combination with iadademstat in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3 (Karnofsky ≥ 30)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (unless elevated due to Gilbert's syndrome, thought to be related to MPN-AP/BP, or due to extrasvascular hemolysis. In these cases conjugated bilirubin should be ≤ 2.0 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Glomerular filtration rate (GFR) ≥60 mL/min/1.73 m^2 by Modification of Diet in Renal Disease (MDRD)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of ASTX727 (35 mg decitabine + 100 mg cedazuridine) and/or iadademstat on the developing human fetus are unknown. For this reason and because DNMT inhibitor and LSD1 inhibitor agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and 6 months after completion of ASTX727 (35 mg decitabine + 100 mg cedazuridine) and/or iadademstat administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation and 6 months after completion of ASTX727 (35 mg decitabine + 100 mg cedazuridine) and/or iadademstat administration
* Women of child-bearing potential must agree not to donate or freeze egg(s) during the course of this study or within 180 days after receiving their last dose of study drug. Male patients must agree not to donate sperm during the course of this study or within 180 days after receiving their last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Patient is able to swallow oral medications
* Patients must have a body weight of at least 50 kg due to the use of flat doses. If a patient is on continued treatment and is receiving benefit, but falls below 50 kg, they may stay on the study per investigator discretion. Otherwise, they will have to come off the study
* Peripheral white blood cell (WBC) count <25 x 10^9/L on day 1 prior to treatment initiation. Hydroxyurea is allowed for cytoreduction until 24 hours prior to study treatment

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents or had received any investigational products within 3 weeks or 5 half-lives (whichever is shorter) prior to first dose of study treatment
* Patients with a QTcF > 450 ms
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASTX727 (35 mg decitabine + 100 mg cedazuridine) or iadademstat
* Patients medicated with anti-depressants reported to have KDM1A/LSD1 inhibitory activity: tranylcypromine or phenelzine
* Patients with IDH1-mutated MPN blast phase (≥20% blasts). Patients with an IDH1-mutation with MPN-AP (10-19%) blasts are eligible for this study
* Iadademstat concomitant medication considerations: Patients are not allowed to receive prophylactic hematopoietic colony stimulating factors, any complementary or alternative medicine [any of various systems of healing or treating disease (as non-prescription supplements, herbal medicine and homeopathy)]. Of note, patients may receive granulocyte colony-stimulating factor for management of febrile neutropenia or for prolonged neutropenia
* Patients may not receive administration of live or live-attenuated vaccines. Administration of non-live vaccines included ribonucleic acid (RNA)-based vaccines is allowed and is recommended for pneumococcal, coronavirus, and influenza vaccines
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because iadademstat is an LSD1 inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with iadademstat, breastfeeding should be discontinued if the mother is treated with iadademstat. These potential risks also apply to the ASTX727 (35 mg decitabine + 100 mg cedazuridine) used in this study
* Patients who require treatment while on study with concomitant drugs that target the 5HT2B receptor or the sigma nonspecific receptor (e.g., escitalopram, fluoxetine, sertraline) except for drugs that are considered absolutely essential for the care of the patient and with appropriate treatment monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute leukemia response-complete (ALR-C) rate | Within 4 cycles (cycle length = 28 days)
  ALR-C rates will be compared between the two treatment arms using Fisher's exact test at the one-sided, alpha = 0.15 significance level.

SECONDARY OUTCOMES:
Event-free survival | From day 1 of randomization to the date of treatment failure, hematological relapse from ALR-C, or death from any cause up to 2 years
  Treatment failure is defined as not achieving ALR-C by four cycles of therapy. Hematological relapse is defined as ≥ 5% blasts in bone marrow or peripheral blood or development of myeloid sarcoma after achievement of ALR-C or better. Kaplan-Meier curves will be generated and the two treatment arms will be compared using a stratified log rank test. Cox regression modeling, including treatment arm and dichotomized blast percentage as covariates, will also be performed to estimate the hazard ratio, along with a 90% confidence interval.
Overall survival (OS) | From randomization to the time of death due to any cause up to 2 years
  Kaplan-Meier curves will be generated, and the two treatment arms will be compared using a stratified log rank test. Cox regression modeling including treatment arm and dichotomized blast percentage as covariates, will also be performed to estimate the hazard ratio, along with a 90% confidence interval.
Percentage of allogeneic hematopoietic stem cell transplantation (allo-HCT) | Up to 2 years
  Descriptive statistics will be utilized for analysis and will be broken down by which treatment arm to which a patient is assigned. The number receiving allo-HCT will be compared between the two treatment arms using Fisher's exact test.

OTHER OUTCOMES:
Gene expression levels | After one cycle of therapy (cycle length = 28 days)
  Will be compared between the two treatment groups using two-sample t-tests following log2 transformation.
Transcriptional changes in proliferative pathways and molecular pathways associated with resistance/disease progression | Up to 2 years
  Will be summarized descriptively.
Correspondence between responses | Up to 2 years
  Correspondence between responses as determined by the European LeukemiaNet 2022 acute myeloid leukemia criteria versus the 2012 blast phase myeloproliferative neoplasm criteria will be assessed using McNemar's test.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be described and graded using National Cancer Institute Common Terminology Criteria for Adverse Events. AEs will be summarized by type, severity grade, and attribution to treatment. Comparisons between treatment arms will be performed using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Anand A Patel, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (24):
- United States (24):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm